CLINICAL TRIAL: NCT03063021
Title: A Phase 1 Open Label Dose Ranging Study to Assess the Safety and Tolerability of N-Acetylcysteine (NAC) in Patients With Retinitis Pigmentosa (FIGHT-RP1 Study)
Brief Title: The FIGHT-RP1 Study
Acronym: FIGHT-RP1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00103296
Record Dates: First submitted 2017-02-16; First posted 2017-02-24 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2021-12

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (carbonyl content >0.6, GSH/GSSG <3) (Experimental): Subjects with RP will be enrolled in the experimental arm if they have a high carbonyl content (>0.6) and a reduced GSH/GSSG ratio (<3.0) in the aqueous.
  Interventions: Drug: N-Acetyl Cysteine (NAC)
- Exploratory Arm (carbonyl content <0.6, GSH/GSSG >3) (Experimental): Subjects with RP who don't have a high carbonyl content (>0.6) and a reduced GSH/GSSG ratio (<3.0) but otherwise are good candidates for the study will be enrolled in the exploratory arm.
  Interventions: Drug: N-Acetyl Cysteine (NAC)

INTERVENTIONS:
Drug: N-Acetyl Cysteine (NAC) — Oral tablets of N-acetyl-cysteine

SUMMARY:
Retinitis Pigmentosa (RP) is a devastating eye disease and at present there are no known treatment options that can alter the rate of vision loss. In a series of studies in animal models, the effects of exposing cones in the periphery of the retina to a large excess of oxygen results in progressive oxidative damage to cone photoreceptors and cone cell death. Compared to control patients, those with RP showed significant reduction in the reduced to oxidized glutathione ratio (GSH/GSSG) in aqueous humor and a significant increase in protein carbonyl content. This demonstration of oxidative stress and oxidative damage in the eyes of patients with RP, suggests that oxidative damage-induced cone cell death in animal models of RP may translate to humans with RP and support the hypotheses that (1) potent antioxidants will promote cone survival and function in patients with RP and (2) aqueous GSH/GSSG ratio and carbonyl content on proteins provide useful biomarkers of disease activity in this patient population. Orally administered N-Acetylcysteine (NAC) has been found to be a particularly effective antioxidant that promotes prolonged cone survival and maintenance of cone function in a mouse model of RP. There is good rationale to test the effect of NAC in patients with RP. The first step is to test different dosing regimens to identify the lowest dose that is able to restore aqueous GSH/GSSG ratio and reduce carbonyl adducts on aqueous proteins.

In patients with Idiopathic Pulmonary Fibrosis, polymorphisms within the TOLLIP gene were found to influence outcomes of NAC-treated patients. The product of the TOLLIP gene, toll-interacting protein, is an inhibitory adaptor protein downstream of toll-like receptors, mediators of innate and adaptive immunity. The identification of the influence of TOLLIP polymorphisms on the effect of NAC in Idiopathic Pulmonary Fibrosis provides the rationale for collecting DNA and genotyping the same single nucleotide polymorphisms (SNPs) in the current trial. In addition to this candidate gene genetic analysis, patient RNA will be collected and banked for future transcriptome analysis. The rationale for this is to identify gene expression changes that modify disease progression in RP. There is substantial variability in the rate of progression among patients with RP. A patient who loses all vision early in life can have a sibling with the same mutation who maintains vision into advanced age. This suggests that modifier genes can have a major impact on cone survival. This study will test the hypothesis that the level of expression of gene products that contribute to the antioxidant defense system may influence cone cell death and hence the rate of loss of visual field. It is also possible that gene expression differences may contribute to differences in response to NAC. For these reasons collecting RNA samples from patients will allow next-generation sequencing in the future to understand the transcriptome background on which the study intervention has been performed.

ELIGIBILITY:
Inclusion Criteria:

All subjects must meet the following criteria to be eligible for study entry:

* Signed informed consent and authorization of use and disclosure of protected health information
* Age >18 years
* Patients diagnosed with RP by the investigators, based on clinical phenotype and diagnostic tests

Exclusion Criteria:

Subjects who meet any of the following criteria will be ineligible for study entry:

* Patients with concurrent retinal pathologies that result in vision loss, including but not limited to retinal vein occlusion, diabetic retinopathy and neovascular age-related macular degeneration. If one eye does not have any retinal pathology other than RP, it may be enrolled in the study.
* Patients with uncontrolled arterial hypertension defined as diastolic blood pressure > 95 mm Hg or systolic blood pressure > 160 mm Hg despite medical therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Assessment of safety and tolerability of N-Acetylcysteine including incidence and severity of systemic and ocular adverse events (AEs) and changes from baseline vital signs and physical examination. | Up to 10 months
  Assessment of safety and tolerability of N-Acetylcysteine including incidence and severity of systemic and ocular adverse events (AEs) and changes from baseline vital signs and physical examination.

SECONDARY OUTCOMES:
Change from baseline aqueous and serum carbonyl content and GSH/GSSG ratio at 1 month after initiation of N-Acetylcysteine . | 1 month after initiation of N-Acetylcysteine
Change from baseline aqueous and serum carbonyl content and GSH/GSSG ratio at 2 months after initiation of N-Acetylcysteine . | 2 months after initiation of N-Acetylcysteine
Change from baseline aqueous and serum carbonyl content and GSH/GSSG ratio at 3 months after initiation of N-Acetylcysteine . | 3 months after initiation of N-Acetylcysteine
Change from baseline aqueous and serum carbonyl content and GSH/GSSG ratio at 4 months after initiation of N-Acetylcysteine . | 4 months after initiation of N-Acetylcysteine
Change from baseline aqueous and serum carbonyl content and GSH/GSSG ratio at 5 months after initiation of N-Acetylcysteine . | 5 months after initiation of N-Acetylcysteine
Change from baseline aqueous and serum carbonyl content and GSH/GSSG ratio at 6 months after initiation of N-Acetylcysteine . | 6 months after initiation of N-Acetylcysteine
Change from baseline aqueous and serum carbonyl content and GSH/GSSG ratio at 7 months after initiation of N-Acetylcysteine . | 7 months after initiation of N-Acetylcysteine
Change from baseline aqueous and serum carbonyl content and GSH/GSSG ratio at 8 months after initiation of N-Acetylcysteine . | 8 months after initiation of N-Acetylcysteine
Change from baseline aqueous and serum carbonyl content and GSH/GSSG ratio at 9 months after initiation of N-Acetylcysteine . | 9 months after initiation of N-Acetylcysteine
Change from baseline best corrected visual acuity (BCVA) 6 months after initiation of N-Acetylcysteine | 6 months after initiation of N-Acetylcysteine
Change from baseline central retinal sensitivity by microperimetry 3 months after initiation of N-Acetylcysteine | 3 months after initiation of N-Acetylcysteine
Change from baseline central retinal sensitivity by microperimetry 6 months after initiation of N-Acetylcysteine | 6 months after initiation of N-Acetylcysteine
Change from baseline central retinal sensitivity by microperimetry 9 months after initiation of N-Acetylcysteine | 9 months after initiation of N-Acetylcysteine
Change from baseline ellipsoid zone (EZ) width by spectral domain optical coherence tomography (SD-OCT) 6 months after initiation of N-Acetylcysteine | 6 months after initiation of N-Acetylcysteine
Change from baseline aqueous levels of N-Acetylcysteine | 1, 2, 3, 4, 5, 6, 7, 8, and 9 months after initiation of N-Acetylcysteine
Change from baseline plasma levels of N-Acetylcysteine | 3 and 6 months after initiation of N-Acetylcysteine

CONTACTS AND LOCATIONS:
Locations (1):
- Wilmer Eye Institute, Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Campochiaro PA, Iftikhar M, Hafiz G, Akhlaq A, Tsai G, Wehling D, Lu L, Wall GM, Singh MS, Kong X. Oral N-acetylcysteine improves cone function in retinitis pigmentosa patients in phase I trial. J Clin Invest. 2020 Mar 2;130(3):1527-1541. doi: 10.1172/JCI132990. PMID 31805012

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT03063021/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/21/NCT03063021/ICF_001.pdf